CLINICAL TRIAL: NCT01770457
Title: Cytokine Response in Septic Shock
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Anand Kumar, Attending physician/ investigator WRHA, University of Manitoba
Other Study IDs: B2009:130
Record Dates: First submitted 2013-01-15; First posted 2013-01-17 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: Septic Shock
Keywords: ICU population
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum samples will be collected at specific time points. Initial time point determined by start of Vasopressors Then sequential serum samples will be drawn from patients to examine a broad range of cytokine responses (TNF, IL-1, IL-6, MIF, LIF, HMGB1, etc)
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is designed to examine the early sequential cytokine responses during antibiotic therapy and resuscitation of septic shock in relation to clinical manifestations of disease.

The specific objective is to obtain sequential serum samples from patients with septic shock, examine a broad range of cytokine responses (TNF, IL-1, IL-6, MIF, LIF, HMGB1, etc) in a rigorous manner and correlate these responses to administration of antibiotics, resuscitative efforts and physiologic responses to illness (temp, HR, blood pressure, WBC, etc).

DETAILED DESCRIPTION:
Patients must be on vasopressors Patients cannot be on pressors for > 24 hrs prior to consent

ELIGIBILITY:
Inclusion Criteria:

* Adult ICU patients: . 18 years admitted with septic shock
* Receiving Vasopressors < 24 hrs

Exclusion Criteria:

* Consent refused by patient or SDM
* Received Vasopressors > 24hrs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients with septic shock admitted to intensive care units who are receiving vasopressors for septic shock for <24 hrs. No significant exclusions exist.
Sampling Method: Non-Probability Sample
Enrollment: 325 (Estimated)
Dates: Start 2006-04; Primary Completion 2014-02 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Cytokine response in septic shock | Hours 0, 3, 6, 12, 18, 24, 36, 48, 96 and day 7
  his study is designed to examine the early sequential cytokine responses during antibiotic therapy and resuscitation of septic shock in relation to clinical manifestations of disease.
  The specific objective is to obtain sequential serum samples from patients with septic shock, examine a broad range of cytokine responses (TNF, IL-1, IL-6, MIF, LIF, HMGB1, etc) in a rigorous manner and correlate these responses to administration of antibiotics, resuscitative efforts and physiologic responses to illness (temp, HR, blood pressure, WBC, etc).

CONTACTS AND LOCATIONS:
Overall Officials: Anand Kumar, MD, Principal Investigator — University of Manitoba
Locations (1):
- Health Sciences Centre, Winnipeg, Winnipeg, Manitoba, Canada